CLINICAL TRIAL: NCT01100632
Title: Effectiveness Evaluation of Panax Ginseng, Vitamins and Minerals in Improvement of Stress and Fatigue
Status: Suspended | Phase: Phase 3 | Type: Interventional
Sponsor: Azidus Brasil (Industry)
Responsible Party: Alexandre Frederico, LAL Clinica Pesquisa e Desenvolvimento Ltda
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GEREMS0310; Version 01 - March 11, 2010
Record Dates: First submitted 2010-04-07; First posted 2010-04-09 (Estimated); Last update posted 2010-10-27 (Estimated); Status verified 2010-04

CONDITIONS: Reduction of Stress and Fatigue
MeSH Terms: conditions — Fatigue | interventions — Asian ginseng; Vitamins; Minerals

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Treatment (Experimental): Treatment with the combination of Panax ginseng, vitamins and minerals
  Interventions: Dietary Supplement: Ginseng, vitamins, minerals
- Placebo (Placebo Comparator): Placebo.
  Interventions: Other: Placebo - Gelatin capsule

INTERVENTIONS:
Dietary Supplement: Ginseng, vitamins, minerals — 2 capsules per day
  Arms: Treatment
Other: Placebo - Gelatin capsule — 2 capsules per day
  Arms: Placebo

SUMMARY:
We hope that with the drug, patients obtain reduced levels of stress and fatigue, according to the scales that we use in the study. Hopefully the results of the treated group are significantly higher than the control group (placebo).

ELIGIBILITY:
Inclusion Criteria:

* Agree with all study procedures, signing the IC in two ways;
* Patients older than 18 years, male or female, regardless of ethnicity or social class;
* Presence of mild to moderate stress, confirmed with the Stress Symptom Inventory (ISS);
* Presence of staff fatigue with a score greater than 36 according to the Fatigue Severity Scale (FSS).

Exclusion Criteria:

Constitute exclusion criteria of the study:

* Participation in clinical trials in the 12 months preceding the survey;
* Current treatment with drugs that are stimulants or central nervous system depressants such as hypnotics, anxiolytics, antipsychotics, antidepressants, statins and muscle relaxants;
* Alternative therapies that scientifically, or have no influence in the tables of stress or fatigue as color therapy, acupuncture or relaxing massages;
* Treatment psychotherapeutic medication or not;
* Current treatment or prediction of treatment with oral anticoagulants (due to interaction with the tocopherol);
* Women who are pregnant or lactating;
* Patients with lactose intolerance;
* Patients allergic to soy or peanuts;
* chronic renal failure;
* Patients using other multivitamins or individual vitamins such as vitamin D and / or A.
* Chronic alcoholism;
* Patients with clinical diagnosis of diseases causing severe chronic pain or adversely affect the clinical interpretation as fibromyalgia, multiple sclerosis, neuropathies and myopathies;
* Patients with hypothyroidism or hyperthyreosis diagnosed clinically;
* Patient history and physical examination suggestive of severe hepatorenal failure;
* Patients with decompensated diabetes mellitus (fasting glucose above 180 mg / dL);
* Patients undergoing treatment for cancer;
* Amendment of the routine of life during the study as early vacation or suspected change in working hours;
* Patients with complaints of excessive sleepiness caused by organic disease such as sleep apnea and morbid obesity (BMI above 35);
* History of hypersensitivity to any component of the product under investigation;
* Any finding of clinical observation (clinical history or physical examination) that is interpreted by the physician investigator as a risk to the patient's participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2010-09; Primary Completion 2010-11 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Reduction of stress and fatigue | 14 and 28 days
  1. Stress: ISS Scale will be assessed by the scale - Inventory of Symptoms of Stress in the time selection / screening, 14 and 28 days ± 2 days of treatment.
  2. Fatigue: FSS Scale will be assessed by the scale - Fatigue Severity Scale Selection in The Times / Triage, 14 and 28 days ± 2 days of treatment.

SECONDARY OUTCOMES:
Quality of life and Sexual Function | 14 and 28 days
  c) Quality of life: the quality of life of patients will be assessed using the Short Form 36 questionnaire (SF-36) during the period included 14 and 28 days ± 2 days of treatment.
  d) Sexual function: evaluation of possible changes in libido or sexual performance that this drug will develop will be made by direct questioning by the doctor to the patient inclusion period 14 and 28 days ± 2 days of treatment.